CLINICAL TRIAL: NCT04596085
Title: A Double Blind, Randomized, Placebo Controlled Study to Evaluate Efficacy and Safety of "VIRACIDE" in the Management of Corona Virus Disease 2019 (COVID-19)
Brief Title: Study to Evaluate Efficacy and Safety of "VIRACIDE" IN THE MANAGEMENT OF CORONA VIRUS DISEASE 2019 (COVID-19)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Herb, Inc (Industry)
Collaborators: ProRelix Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NS-VC-CT01-20
Record Dates: First submitted 2020-10-19; First posted 2020-10-22 (Actual); Results first posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Covid19
Keywords: Coronavirus, (SARS-CoV-2)
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: Double Blind, Randomized, Placebo Controlled
Who Masked: Participant, Investigator
Masking Description: Randomized, Double - Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational product (Active Comparator): Experimental, Investigational Product Ingredient : ViraCide Dosage form softgels . Fequency: 3 soft gels, two times every day after breakfast and dinner . Duration: 14 days+ SOC Therapy
  Interventions: Dietary Supplement: Investigational Product - ViraCide
- Placebo (Placebo Comparator): Ingredient, Placebo Ingredient Starch softgels. Frequency: 3 soft gels, two times everyday after breakfast and dinner . Duration:14 days + SOC Therapy
  Interventions: Other: Placebo - Starch Powder Soft gels

INTERVENTIONS:
Dietary Supplement: Investigational Product - ViraCide — Viracide
  Other Names: Investigational Product
  Arms: Investigational product
Other: Placebo - Starch Powder Soft gels — Starch Powder Soft gels
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This is a double blind randomized placebo controlled study will be conducted on 124 subjects, 50 years and older with mild or asymptomatic COVID-19. If symptomatic, symptoms are mild (cough, weakness, sore throat, low grade fever 38.50С, respiratory rate should not be more than 22 / min, resting SpO2 >95%, normal highly sensitive C-reactive protein (HS-CRP) (<10mg/L). There are no signs of dehydration, sepsis or shortness of breath.

The study will be conducted at two centers. There will be a screening visit at Day -4 followed by three visits at the center at Days 1, 7 and 15 and a follow-up visit on Day 28. All participants will be randomized to receive either ViraCide (investigational product) or matching placebo. All subjects will receive SOC therapy.

Note: If subject is discharged before Day 15 PI's discretion as per patients health condition, then assessments scheduled for Day 15 will be carried out on the discharge day (as far as possible and those not performed will be noted on appropriate CRF page) and Day 15 visit will be done telephonically.

DETAILED DESCRIPTION:
Day 1 Randomization, Vital Signs, Pulse oximetry, AE/SAE, Concomitant Medication, ViraCide/ Placebo treatment start, NEWS scoring; 7-point ordinal scoring Day 7 Physical Examination, Vital Signs, AE/SAE, Concomitant Medication, ViraCide/ Placebo Compliance check, Pulse oximetry; NEWS scoring; 7-point ordinal scoring.

(Note: If the subject is discharged on this day as per PI's discretion and patient's health condition then assessment scheduled for day 15 will be carried out on discharge day).

Day 15 Physical Examination, Vital Signs, AE/SAE, Concomitant Medication, ViraCide/ Placebo treatment end, RT-PCR for Sars- Co-V2, Hs-CRP, Safety Lab Tests, Pulse oximetry; NEWS scoring; 7-point ordinal scoring, ViraCide/ Placebo Compliance check, Lab assessment including urine analysis Day 28

Phone call follow up for time :

* until negative RT-PCR for Sars-Co- V2, COVID-19 related mortality,
* development of any COVID-19 symptom,
* development of any worsening of comorbid condition;
* Development of new AE/SAE; Resolution status of previous AE/SAEs

Note: If subject is discharged before Day 15on PI's discretion as per patients health condition, then assessments scheduled for Day 15 will be carried out on the discharge day (as far as possible and those not performed will be noted on appropriate CRF page) and Day 15 visit will be done telephonically.

ELIGIBILITY:
Inclusion Criteria:

1. 50 years or older
2. Both male and female subjects will be included
3. Positive oropharyngeal/nasal swab RT-PCR for Sars-Co- V2. Diagnosed not more than 2 days ago(diagnosis

   ≤2days).
4. Either asymptomatic or have mild symptoms. Onset of symptoms within no more than 4 days If symptomatic, symptoms are mild (cough, weakness, sore throat, low grade fever 38.50С, respiratory rate should not be more than 22 / min, resting SpO2 >95%, normal highly sensitive C-reactive protein (HS-CRP) (<10mg/L). There are no signs of dehydration, sepsis or shortness of breath.
5. Chronic stable medical conditions: diabetes mellitus, or hypertension, or chronic heart disease. Under treatment and controlled by medication
6. Signed informed consent/or consent given through text message, WhatsApp ore-mail.
7. Ability to understand the requirements of the Research Protocol and follow the research procedures.
8. Subject should be willing to be managed in isolation wards
9. Negative pregnancy test (for female participants)
10. Adequate contraception for study duration

Exclusion Criteria:

1. Less than 50years
2. With severe COVID-19 symptoms requiring immediate hospitalization
3. Investigator considers the subject unsuitable for ViraCide
4. History of symptoms of more than 4days
5. COVID-19 diagnosed >2 days ago using oropharyngeal/nasal swab RT-PCR forSars-Co-V2
6. History of cardiopulmonary resuscitation
7. Subjects having history of organ failure or conditions requiring ICU monitoring and treatment, such as severe liver disease, severe renal dysfunction, upper gastrointestinal hemorrhage, disseminated intravascular coagulation or any other condition that in the PI"s opinion makes the subject unfit to participate
8. Respiratory failure, ARDS or need of mechanical ventilation
9. History of acute exacerbation of comorbidity like heart failure, diabetic ketoacidosis, myocardial infection, major cardiac rhythm disorder or any other condition that in the PI"s opinion makes the subject unfit to participate
10. History of or current hepatic failure or severely compromised liver function, or renal failure or having chronic kidney disease or acute renal failure
11. History of or currently receiving treatment for an endocrine disorder like hypothyroidism, hyperthyroidism that is likely to affect the basal heart rate.
12. History of or currently under treatment for asthma [exception: patients with history of asthma, not on medications/inhalers/nebulizers for at least 6 months before study start), COPD, bronchiectasis, asbestosis and other such chronic lung conditions that can compromise SpO2 and RR.
13. HIV, HBsAg, HCV positive
14. Any condition causing immunodeficiency
15. Systemic connective tissue disease or any autoimmune disease that is likely to affect HS-CRP levels
16. History of epilepsy/epileptic fit/convulsions in last 6 months or currently on treatment for it
17. History of or currently having malignancy and being treated for it. (exception: histologically confirmed and cured carcinoma in situ)
18. Hypersensitivity reaction to Study drug/placebo
19. Any psychiatric issue for which the subject is currently undergoing treatment
20. Any history of drug/alcohol dependence within 30 days of screening or current drug/alcohol dependence
21. Inability to understand the requirements of the Research Protocol and follow the research procedures.
22. Pregnant or lactating;
23. Not willing to use adequate contraception during study duration
24. Participation in any other clinical study less than 3months before the start of the study.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2020-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Ninad Naik, MD(Ayurveda), Principal Investigator — Gunjkar Multispeciality Hospital; Dr. A Gopal Rao, MD(Med), Principal Investigator — Government medical college and Government general hospital
Locations (2):
- India (2):
  - Department of General medicine/ clinical research. Government medical college and Government general hospital, Srikakulam, Andhra Pradesh
  - Gunjkar Multispeciality Hospital, Pune, Maharashtra

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Investigational Product | Placebo
Started | 59 | 59
Completed | 59 | 59
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational Product | Placebo | Total
Number analyzed (Participants) | 59 | 59 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.53 (5.81) | 60.44 (7.01) | 59.48 (6.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 38 | 36 | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 59 | 59 | 118
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With National Early Warning Score (NEWS) Change From 3 to 0
Description: The proportion of cases with National Early Warning Score reduction from 3 to 0 till discharge day between two groups.
  This score is associated with clinical risk and a decrease in score indicates a decrease in the risk to the patient and improvement in clinical condition.
Time Frame: First treatment date up to discharge day, an average of 1 week
Measure: Count of Participants; unit: Participants
Groups:
- Investigational Product: Experimental, Investigational Product Ingredient : ViraCide Dosage form softgels .
- Placebo: Ingredient, Placebo Ingredient Starch softgels.
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 59 | 59
Participants | 44 | 29

2. Primary Outcome: Number of Participants With 7-point Ordinal Scale Score Change From 3 to 1
Description: Proportion of cases with 7-point ordinal scale score reduction from 3 to 1 till day 7.
  This score is associated with clinical improvement and a decrease in score indicates improvement in patient's clinical condition.
Time Frame: First treatment date up to day 7, i.e. up to 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 59 | 59
Participants | 45 | 28

3. Primary Outcome: Time to a Negative COVID-19 Nucleic Acid Testing
Description: Time to COVID-19 nucleic acid testing negativity in oropharyngeal/nasal swab)
Time Frame: Time Frame: First treatment date up to 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 59 | 59
days | 5.47 (0.49) | 6.97 (0.61)

4. Primary Outcome: Rate of Progression on National Early Warning Score
Description: Rate of progression to the severe/critical COVID-19 disease
Time Frame: First treatment date up tp 28 days (28 days)
Population: The Rate of progression to the severity of the disease was not identifiable as most of the subjects were discharged on Day 7 or 8
Groups:
- Investigational Product: Experimental, Investigational Product Ingredient : ViraCide softgels . Frequency: 3 soft gels, two times every day after breakfast and dinner.
- Placebo: Ingredient, Placebo Ingredient Starch softgels. Frequency: 3 soft gels, two times every day after breakfast and dinner.
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Rate of Progression on 7- Point Ordinal Scale
Description: Rate of progression to the severe/critical COVID-19 disease
Time Frame: First treatment date up to 28 days
Population: as for outcome 4
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: ICU Admissions
Description: Incidence of ICU admissions
Time Frame: Time frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 59 | 59
Participants | 0 | 0

7. Secondary Outcome: Subject Survival
Description: Subject survival in the trial
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 59 | 59
Participants | 59 | 59

8. Secondary Outcome: Incidence of Mechanical Ventilation
Description: Number of incidences of mechanical ventilation due to COVID-19 infection
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 59 | 59
Participants | 0 | 0

9. Secondary Outcome: Change in Clinical or Laboratory Assessment of Comorbid Condition
Description: To evaluate any decline in health condition due to comorbidity
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 59 | 59
Participants | 0 | 0

10. Secondary Outcome: Percent of Participants With Worsening Comorbid Condition
Description: Percent of participants with worsening comorbid condition.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 59 | 59
percentage | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Investigational Product | Placebo
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 3/59 | 4/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Product (N=59) | Placebo (N=59)
nausea (General disorders) | 1 (1) | 2 (2)
mouth ulcer (General disorders) | 1 (1) | 2 (2)
vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Confidential information during the course of the study and clinical development plan, except the information already existing in the public domain, and all results and reports obtained, collected, conceived, processed and developed pursuant to this Agreement, The INSTITUTION shall use confidential information for the sole purpose of providing services under this Agreement and shall not use confidential information for the INSTITUTION's own benefit at any time.

DOCUMENTS (2):
  • Study Protocol (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT04596085/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/85/NCT04596085/SAP_001.pdf